CLINICAL TRIAL: NCT03090165
Title: A Phase I/II, Single Arm, Non-randomized Study of Ribociclib (LEE011), a CDK 4/6 Inhibitor, in Combination With Bicalutamide, an Androgen Receptor (AR) Inhibitor, in Advanced AR+ Triple-negative Breast Cancer: Big Ten Cancer Research Consortium BRE15-024
Brief Title: Ribociclib and Bicalutamide in AR+ TNBC
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kari Wisinski (Other)
Collaborators: Novartis (Industry); Big Ten Cancer Research Consortium (Other); University of Wisconsin, Madison (Other)
Responsible Party: Sponsor-Investigator, Kari Wisinski, Sponsor Investigator, Big Ten Cancer Research Consortium
Organization: Big Ten Cancer Research Consortium (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTCRC BRE15-024
Record Dates: First submitted 2017-03-01; First posted 2017-03-24 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Triple Negative Breast Cancer
Keywords: Triple Negative Breast Neoplasms; ribociclib; LEE011; CDK 4/6 inhibitor; bicalutamide
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — ribociclib; bicalutamide

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm A - Phase I (Experimental): Dose Escalation Cohort 1 will consist of 3-6 patients who will receive bicalutamide 150mg PO daily on days 1-28 of a 28 day cycle and ribociclib 400mg PO daily on days 1-21 of a 28 day cycle.
  Cohort 2 will consist of 3-6 patients who will receive bicalutamide 150mg PO daily on days 1-28 of a 28 day cycle and ribociclib 400mg PO daily on days 1-28 of a 28 day cycle.
  Cohort 3 will consist of 3-6 patients who will receive bicalutamide 150mg PO daily on days 1-28 of a 28 day cycle and ribociclib 600mg PO daily on days 1-21 of a 28 day cycle.
  Experimental: Arm B - Phase II Investigational Treatment The maximum safe dose of ribociclib in combination with bicalutamide will be given to up to 25 patients.
  Interventions: Drug: ribociclib; Drug: Bicalutamide

INTERVENTIONS:
Drug: ribociclib — 400mg PO
  Other Names: LEE011
Drug: ribociclib — 600mg PO
  Other Names: LEE011
Drug: Bicalutamide — 150mg PO

SUMMARY:
This is an open label, multi-institutional, single arm phase II trial of ribociclib in combination with bicalutamide in advanced AR+ triple-negative breast cancer. No randomization or blinding is involved.

DETAILED DESCRIPTION:
This is a non-randomized, single arm, open label study of the combination of bicalutamide with ribociclib in subjects with advanced AR+ TNBC. Prior to enrollment on the phase II cohort, a phase I run-in study will be performed to ensure safety and tolerability of the combination of bicalutamide and ribociclib in subjects with advanced AR+ TNBC.

In both the phase I and phase II portions of the study, subjects will receive bicalutamide 150 mg orally, once daily, continuously on Day 1 to Day 28. Each cycle of treatment is 28 days.

In the phase I portion of the study, cohorts of subjects will receive ribociclib in escalated doses orally, once daily in a 28 day cycle. For the phase II portion, the RP2D dose of ribociclib will be based on the phase I run-in.

In the phase II cohort, a two week lead-in of bicalutamide monotherapy will occur before cycle 1 combination therapy (Day -14 to day -1). Then ribociclib will be added on day 1 of cycle 1. This lead-in will be for CTC androgen receptor analysis.

ELIGIBILITY:
Individuals from populations who are underrepresented in clinical research (e.g., racial and ethnic minorities, women, individuals from rural/frontier communities, older individuals) will be enrolled with a goal of ensuring that all eligible patients are given the opportunity to participate in novel clinical trials and that research findings can be generalizable to the entire population.

Androgen Receptor (AR) positivity definitions -Phase I: Metastatic or unresectable AR+ triple-negative breast cancer (TNBC); AR positivity defined as IHC staining of >0% of tumor nuclei.

OR

-Phase II: Metastatic or unresectable AR+ triple-negative breast cancer (TNBC); AR positivity defined as IHC staining of ≥10% of tumor nuclei.

Inclusion Criteria for Phase I and II study.

In addition to being AR positive as defined in protocol, subjects must also meet all of the following applicable inclusion criteria.

* Histological or cytological confirmed, metastatic or unresectable triple-negative breast cancer (TNBC). TNBC will be defined as expression of ER<10%, PR< 10% and HER2 negative either by IHC (0, 1+ are negative, 2+ equivocal) or in situ hybridization method (ratio <2.0 is negative).
* Written informed consent and HIPAA authorization for release of personal health information. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
* Up to 3 prior line of systemic therapy for metastatic disease is allowed. Combination therapy will be considered 1 line.
* Age ≥ 18 years at the time of consent.
* ECOG Performance Status of 0, 1 or 2 within 28 days prior to registration.
* Life expectancy of > 12 weeks as determined by the treating physician.
* Measurable disease according to RECIST 1.1 within 28 days prior to registration.
* No active central nervous system (CNS) metastatic disease. NOTE: Subjects with CNS involvement must meet ALL of the following to be eligible:

  * At least 28 days from prior definitive treatment of their CNS disease by surgical resection, stereotactic body radiation therapy (SBRT) or whole brain radiation treatment (WBRT) at the time of registration
  * AND asymptomatic and off systemic corticosteroids and/or enzyme-inducing anti-epileptic medications for brain metastases for >14 days prior to registration.
* Prior cancer treatment must be completed at least 14 days prior to registration and the subject must have recovered from all reversible acute toxic effects of the regimen (other than alopecia) to ≤grade 1 or to baseline prior to initiation of that therapy.
* Screening rate-corrected QT interval (QTc) must be <450msec and a resting heart rate of at least 50-90 bpm via a standard 12-lead ECG within 28 days prior to registration.
* Demonstrate adequate bone marrow and organ function as defined in the protocol; all screening labs to be obtained within 28 days prior to registration.
* Females of childbearing potential must have a negative serum pregnancy test within 7 days prior to registration. NOTE: Females are considered of child bearing potential unless they are surgically sterile (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy), or they are naturally postmenopausal for at least 12 consecutive months, or her male partner has had a vasectomy at least 6 months prior to screening (The sterilized male partner must be her only sexual partner.).
* Females of childbearing potential and males must be willing to abstain from heterosexual activity or must agree to use adequate contraception (hormonal or barrier method) for the duration of study participation and for 3 weeks after discontinuation of study treatment.
* As determined by the enrolling physician or protocol designee, ability of the subject to understand and comply with study procedures for the entire length of the study.
* Able to swallow bicalutamide and ribociclib tablets.

Exclusion Criteria:

* Prior therapy with AR antagonists including but not limited to bicalutamide, enzalutamide, abiraterone and orteronel.
* Prior therapy with any CDK 4/6 inhibitors with the exception of participation in a window or preoperative study for Stage I-III operable breast cancer..
* Active infection requiring systemic therapy.
* Pregnant or breastfeeding (NOTE: breast milk cannot be stored for future use while the mother is being treated on study).
* Known additional malignancy that is active and/or progressive requiring treatment; exceptions include basal cell or squamous cell skin cancer, in situ cervical or bladder cancer, or other cancer for which the subject has been disease-free for at least three years.
* Treatment with any investigational drug within 14 days prior to registration or within 5 half-lives of the investigational product, whichever is longer. Immunotherapies such as PD-L1 or PD-1 inhibitors only require a 14 day window, regardless of half-life. Investigational imaging agents are not included in this definition and are allowed.
* Subject who has received radiotherapy <14 days prior to registration, and who has not recovered to grade 1 or better from related side effects of such therapy (exceptions include alopecia and any adverse events deemed by the investigator to be unlikely to interfere with the study drug safety).
* Subject has had major surgery within 14 days prior to registration or has not recovered from major side effects of the surgery (tumor biopsy is not considered as major surgery).
* Known hypersensitivity to any of the excipients of ribociclib or bicalutamide.
* Any impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of the study drugs (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection).
* Known history of HIV infection (testing not mandatory).
* Any concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgment, cause unacceptable safety risks, contraindicate subject participation in the clinical study or compromise compliance with the protocol (e.g. chronic pancreatitis, chronic active hepatitis, active untreated or uncontrolled fungal, bacterial or viral infections, etc.).
* Subjects with any of the following conditions are excluded:

  * Serious or non-healing wound, ulcer, or bone fracture.
  * History of abdominal fistula, gastrointestinal perforation, or intra- abdominal abscess within 28 days prior to registration.
  * Any history of cerebrovascular accident (CVA) or transient ischemic attack within 12 months prior to registration.
  * Any history of arterial or venous thrombosis/thromboembolic event, including pulmonary embolism within the past 12 months prior to registration.
  * History of acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass grafting, coronary angioplasty, or stenting) or symptomatic pericarditis within 6 months prior to registration.
  * Symptomatic congestive heart failure (New York Heart Association III-IV) or documented current cardiomyopathy with left ventricular ejection fraction (LVEF) <50%
  * Clinically significant cardiac arrhythmias (e.g. ventricular tachycardia) or clinically significant, complete left bundle branch block, high-grade AV block (e.g. bifascicular block, Mobitz type II and third-degree AV block).
  * Any episode of atrial fibrillation in the prior 12 months.
  * Long QT syndrome or family history of idiopathic sudden death or congenital long QT syndrome.
  * Concomitant use of medication(s) with a known risk to prolong the QT interval and/or known to cause Torsades de Pointe that cannot be discontinued (within 5 half-lives or 7 days prior to starting study drug) or replaced by safe alternative medication. See ManualDocuments/Info tab of the EDC for list of medications.
  * Systolic blood pressure (SBP) >160 mmHg or <90 mmHg at screening.
* Currently receiving any known strong inducers or inhibitors of CYP3A4/5 which cannot be discontinued 7 days prior to starting study drug (see Appendix 1 for details).
* Subject is currently receiving or has received systemic corticosteroids <14 days prior to starting study drugs. The following uses of corticosteroids are permitted: a short duration (<5 days) of systemic corticosteroidssingle doses, any duration of topical applications (e.g., for rash), inhaled sprays (e.g., for obstructive airways diseases), eye drops or local injections (e.g., intra-articular).
* Subject is currently receiving warfarin or other coumarin-derived anticoagulant for treatment, prophylaxis or otherwise. Therapy with heparin, low molecular weight heparin (LMWH), novel oral anticoagulants (NOACs) or fondaparinux is allowed.
* In subjects with a diagnosis of cirrhosis, sSubjects with a Child-Pugh score B or C are excluded. Please see chart in the ManualDocuments/Info tab of the electronic data capture system (EDC) for Child-Pugh score calculation. If subject does not have diagnosed or suspected cirrhosis, the Child-Pugh score does not need to be calculated.
* Subjects taking herbal supplements (St. John's Wort, gingko balboa, etc.) must discontinue these supplements 14 days prior to study registration.
* Consumption of grapefruit, grapefruit hybrids, pummelos, star-fruit, Seville oranges or products containing the juice of each within 7 days prior to study registration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2018-05-07 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Phase I: Maximum Tolerated Dose | D1 of treatment to end of cohort cycle (assessed at 28 days)
  Phase I: Maximum tolerated dose (MTD) for subjects receiving ribociclib and bicalutamide without experiencing dose-limiting toxicity(s) (DLT) per Common Terminology Criteria for Adverse Events (CTCAE) v4
Phase II: Clinical benefit rate (CBR) of treatment combination | D1 of treatment to end of 4 treatment cycles (assessed at 16 weeks)
  Compare sum of confirmed complete plus partial responses plus stable disease per response evaluation criteria in solid tumors (RECIST) 1.1 criteria

SECONDARY OUTCOMES:
Phase I: Objective Response Rate (ORR) | 2 years
  The objective response rate is the proportion of all subjects with confirmed PR or CR according to RECIST 1.1, from the start of treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the start of treatment).
Phase I: Duration of Response | 2 years
  Duration of overall response-the period measured from the time that measurement criteria are met for complete or partial response (whichever status is recorded first) until the date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since treatment started).
Phase I: Assess Safety and Tolerability By summarizing counts and percentages grade 3-5 adverse events (NCI CTCAE Version 4) | 2 years
  By summarizing counts and percentages grade 3-5 adverse events (NCI CTCAE Version 4)
Phase I: Ribociclib pharmacokinetics | 2 months
  Time points: Peak Plasma Concentration (Cmax) Pre dose and 2-hours post-dose (±15 min) pharmacokinetic samples will be collected on Cycle 1 Day 1, Cycle 1 Day 15, Cycle 2 Day 1 and Cycle 2 Day 15.
Phase II: Progression Free Survival (PFS) | 2 years
  PFS will be summarized using Kaplan-Meier estimates of the median survival times.
Phase II: Objective Response Rate (ORR) | 2 years
  by RECIST 1.1 on treatment with combination of bicalutamide and ribociclib in advanced AR+ TNBC
Phase II: Overall Survival (OS) | 5 years
  Overall survival is defined by the date of treatment initiation to date of death from any cause.
Phase II: Estimate Duration of Response | 2 years
  On treatment with combination of bicalutamide and ribociclib in advanced Androgen Receptor (AR)+ Triple Negative Breast Cancer (TNBC)
Phase II: Evaluate Safety and Tolerability By summarizing counts and percentages grade 3-5 adverse events (NCI CTCAE Version 4) | 2 years
  By summarizing counts and percentages grade 3-5 adverse events (NCI CTCAE Version 4)

CONTACTS AND LOCATIONS:
Overall Officials: Kari Wisinski, MD, Principal Investigator — University of Wisconsin, Madison
Locations (6):
- United States (6):
  - University of Illinois Cancer Center, Chicago, Illinois
  - Michigan State University, Lansing, Michigan
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - University of Rochester Medical Center, Rochester, New York
  - Penn State Cancer Institute, Hershey, Pennsylvania
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Big Ten Cancer Research Consortium Website — http://www.bigtencrc.org/